CLINICAL TRIAL: NCT03972332
Title: Pain Experience in Individuals With Chronic Low Back Pain: a Cohort Study
Brief Title: Pain Experience in Individuals With Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Versus Arthritis (Other); Nottingham Biomedical Research Centre (Unknown); Muculoskeletal Association of Chartered Physiotherapists (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17112
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Central Sensitisation; Hyperalgesia; Hypersensitivity
MeSH Terms: conditions — Low Back Pain; Hyperalgesia; Hypersensitivity | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sensitised: Participants with sensitisation that significantly deviates from the normal mean as assessed by Quantitative Sensory Testing
  Interventions: Diagnostic Test: Quantitative Sensory Testing
- Non-sensitised: All other participants with sensitisation that is not significantly deviating from the normal mean as assessed by Quantitative Sensory Testing
  Interventions: Diagnostic Test: Quantitative Sensory Testing

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Testing — PPT: An electronic data collection unit will be used featuring an electronic algometer connected with a laptop where the amount of pressure will be displayed on the screen. When the pressure pain detection threshold is reached (the point where the pressure sensation starts to be experienced as pain), the individual will press a button at a handheld device, that will automatically store the pressure value in the system and serve as an indication, for the examiner, to stop the testing.
  TS: A pinprick stimulator (Weight: 256mNewton) will be used. The examiner will apply the pen that features a retractable blunt needle in a repetitive manner (once per second for ten seconds). The individual will be asked for the intensity of pain (NRS) at the first and at the last time and the given score will be noted.
  CPM: A manual blood pressure sphygmomanometer will be used in conjunction with the electronic algometer described above (PPT).
  Other Names: Pain Pressure Detection Threshold (PPT); Temporal Summation (TS); Conditioned Pain Modulation (CPM)

SUMMARY:
Low back pain is a very common musculoskeletal condition that affects many people each year regardless of age, gender, and ethnicity. Most people get better however, some continue suffering from painful episodes despite treatment.

Self-management strategies for the management of chronic low back pain are very important to patients as they help them develop skills to manage their pain more effectively. However, self-management strategies are not always effective as expected. It is possible that the brain has become very sensitive to signals coming from peripheral parts of the body (e.g. low back) affecting the ability of patients to self-manage their condition.

The aim of this study is to establish whether central sensitisation (sensitivity of the brain to peripheral signals) predicts how effective self-management approaches will be.

On three different occasions, scheduled sessions will include a clinical assessment session and completion of a questionnaire booklet. The clinical assessment will measure three features of central sensitisation: 1) sensitivity to blunt pressure on the forearm, 2) changes in pain, felt during repeated light pricking of the forearm skin, and 3) reduction in pain that accompanies inflation of a blood pressure cuff on the opposite arm. Participant involvement at each session is expected to last for 70 minutes.

Individuals over 18, diagnosed with chronic low back pain and enlisted to follow a pain management program are eligible to participate. The clinical assessments, questionnaire completion and subsequent statistical analysis are expected to be completed within 18 months of study commencement.

Based on our findings, future research may use similar clinical assessment to identify people who might be helped to self-manage by using treatment that reduces central sensitisation.

DETAILED DESCRIPTION:
Low Back Pain (LBP) is considered a common condition consisting of a set of complains (pain, muscle tension, or stiffness), manifesting primarily to the lower back region (below the costal margin and above the inferior gluteal folds). LBP may or may not include radiating pain to the lower limb and can be caused by a number of underlying pathologies with varying levels of severity [1]. The condition can be the result of complex interactions between multiple physical and psychological factors including osteoarthritis (OA), degenerated discs, disc herniation, muscle dysfunction, obesity, poor posture, mental illness, negative affect (stress, anxiety, depression) [2].

LBP lifespan incidence appears to be 58-84% while it is estimated that 11% of males and 16% of females suffer from chronic LBP at any point in time [3]. It is expected that 40-50% of individuals suffering from acute LBP will continue to experience pain at three months and will demonstrate little or none further improvement, while 60-70% of those who improve will relapse within a year [4]. The global prevalence of LBP demonstrates continuously growing trends with a 17.3% increase in the last 10 years [5].

Self-management (SM) support is a portfolio of techniques and tools to help patients choose healthy behaviours as well as a fundamental transformation of the patient-caregiver relationship into a collaborative partnership [6]. Self-management support has to incorporate in its approach elements that aim to increase patients' self-efficacy, develop problem-solving, decision-making and goal-setting skills as well as to promote partner-like behaviour between patients and health professionals [7]. SM interventions pose as ideal rehabilitation strategies for chronic low back pain (CLBP) as they aim to address biological (neurophysiological, deconditioning, lifestyle) and psychosocial (self-efficacy, maladaptive beliefs, anxiety/depression) factors that have been identified as risk factors for poor outcome [8, 9] and are negatively affected by central sensitisation (CS) [10]. SM interventions are designed to be cost-effective by reducing health care utilisation associated with LBP [11].

Self-management programs (SMP) for CLBP demonstrate only small to moderate effects for long-term improvements in pain and disability. Currently, it is not known what factors predict effective self-management. Evidence of CS varies between individuals with chronic pain, and may contribute to the relatively poor efficacy of SMPs.

CS is a marker of widespread and centrally augmented pain that refers to those neurophysiological processes that can occur throughout the central nervous system (CNS) distribution, leading to changes in the spinal cord as well as in the brain [12]. The presence of CS increases the complexity of the clinical picture [13] and negatively affects a range of outcomes (e.g. pain, disability, negative affect, quality of life) following treatment [14]. CS is not present within all patients with chronic pain [15] rendering identification of those patients and decision-making for the right management approach even harder [16]. Patients with potential development of CS should receive treatment that address the full biopsychosocial clinical spectrum consisting of cognitive behavioural therapy (CBT) as well as therapeutic pain neuroscience education [17]. Changes in pain mechanisms may explain the moderate levels of evidence for the effectiveness of self-management (SM) interventions in LBP populations [7] as CS has been shown to negatively affect the perception of back pain, pain-related disability and lead to poor physical and mental health-related quality of life as well as to greater levels of depression and anxiety [10].

Quantitative Sensory Testing (QST) is a reliable [18] and valid [19] method to assess for the presence of CS and demonstrates predictive capacity in relation to musculoskeletal (MSK) treatment outcomes [20]. The testing consists of pressure pain threshold (PPT), punctate thresholds, temperature sensitivity, temporal summation (TS) and conditioned pain modulation (CPM) used to quantify noxious or innocuous stimuli within healthy individuals and patients alike [21]. QST has been used, among others, as a screening and assessment tool for sensory abnormalities in patients with pain disorders [21], as well as to assist in the stratification of patients [22] and evaluate the clinical aspects of peripheral and CS [23].

The STarT Back screening tool [24] was developed for individuals of LBP with the aim to identify prognostic indicators that could potentially assist decision making concerning initial treatment options in primary care [25]. Start Back has been formally validated, displaying satisfactory reliability, and has demonstrated that a stratified management approach displays higher health gains for patients with LBP than a non-stratified one [26]. Nevertheless, the tool's predictive performance has not been examined when other biomarkers (CS) are included as prognostic indicators.

Findings from this research will have an impact on differential diagnosis of chronic pain and CS identification as potential prognostic indicators for self-management. The results will assist effective patient subgrouping (stratification) based on CS measurements, aid appropriate self-management approaches in CLBP and potentially other chronic musculoskeletal pain states.

ELIGIBILITY:
Inclusion Criteria:

* have the ability to give informed consent.
* be 18 years old or over
* be diagnosed with chronic LBP
* be enlisted for participation in a self-management program
* be able to speak and understand English as all questionnaires are validated in the English language.

Exclusion Criteria:

* Inability to give informed consent due to cognitive impairment or otherwise
* Inability to understand key aspects of the study due to cognitive impairment or otherwise
* Patients giving history of additional co-morbidities such as cancer, diabetic neuropathies, fractures or other conditions causing greater disability than their back pain.
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with a confirmed diagnosis of CLBP that have been assigned for participation to a self-management program at a clinical or community setting
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Self-management | 3 months
  Self-management will be assessed with the Health Education Impact Questionnaire (heiQ) that measures the ability of a patient to self-manage their condition and features 40 questions that spread across 8 distinct domains (Health Directed Behavior: 4 items; Positive and Active Engagement in Life: 5 items; Self-Monitoring and Insight: 6 items; Constructive Attitudes and Approaches: 5 items; Skill and Technique Acquisition: 4 items; Social Integration and Support: 5 items Health Service Navigation: 5 items; and Emotional Wellbeing: 6 items). Each item is rated with a 4-level scale (Strongly agree to Strongly disagree) and a number (1-4) is allocated that leads to the calculation of a mean. No single value can be produced for heiQ. Rather, each domain must be used individually. The higher the value the best the self-management ability in all domains apart from Emotional Wellbeing where a high value represents a low self-management ability.

SECONDARY OUTCOMES:
Pain Severity: Numerical Rating Scale (NRS) | 3 months
  Pain will be assessed with the Numerical Rating Scale (NRS) where patients will be asked to rate their current pain on a scale from 0 to 10 with 0 indicating no pain and 10 the worst pain imaginable.
Levels of Disability | 3 months
  Disability will be assessed with the Roland-Morris Disability Questionnaire (RMDQ) where patients are asked to tick a box if they agree with 24 statements regarding their ability to perform certain activities (dressing, housework, walking). If the don't agree with the statement (able to perform thoe activities) they need to leave the tick-box blank or unchecked. Every agreement (tick) counts as a point and an absolute value is formed (min: 0, max: 24). The higher the value the higher the disability level.
Patient Quality of Life: EQ-5D-5L questionnaire | 3 months
  Quality of Life will be assessed with the EQ-5D-5L questionnaire. EQ-5D-5L has two components: health state description and evaluation. In the description part, health status is measured in terms of 5 dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using a five-level (5L) scale (no problem to extremely severe). Each dimension can be used for analysis as a categorical variable or combined with the others as a 5-digit value according to responses (example 11231). On a single dimension, a categorical value of 1 signifies no problem and a value of 5 extremely severe problem. Similarly, a combined value of 11111 shows excellent quality of life whereas a value of 55555 shows a severely affected quality of life.
Self-efficacy: Pain Self-efficacy Questionnaire (PSEQ) | 3 months
  Self-efficacy will be assessed with the Pain Self-efficacy Questionnaire (PSEQ) where patients are asked to indicate their levels of confidence with a 0-6 scale (0 indicates not at all confident and 6 extremely confident)on an array of 10 questions. A sum of all responses is calculated (60 being the maximum) for analysis. The higher the value the higher the levels of self-efficacy.
Fatigue | 3 months
  Fatigue will be assessed with the Fatigue Severity Scale (FSS) where patients are asked to indicate their levels of agreement with a 0-7 scale (0 indicates strong disagreement and 7 strong agreement) at 9 questions. A sum of all responses is calculated (63 being the maximum) for analysis. The higher the value the higher the level of fatigue.
  Also, patients are asked to rate their global fatigue on a 0-10 scale with 0 being worst and 10 being normal fatigue. This sub-scale will be used on its own for analysis.
Anxiety | 3 months
  Anxiety will be assessed with the Anxiety part of the Hospital Anxiety and Depression Scale (HADS) where patients are asked to indicate their levels of emotion frequency with a 4-level scale (0-3: 0 indicates never and 3 all the time) at 7 questions. A sum of all responses is calculated (21 being the maximum) for analysis. The higher the value the higher the levels of anxiety.
Depression | 3 months
  Depression will be assessed with the Depression part of the Hospital Anxiety and Depression Scale (HADS) where patients are asked to indicate their levels of emotion frequency with a 4-level scale (0-3: 0 indicates all the time and 3 never) at 7 questions. A sum of all responses is calculated (21 being the maximum) for analysis. The higher the value the higher the levels of depression.
Catastrophization | 3 months
  Catastrophization will be assessed with the Pain Catastrophizing Scale (PCS) where patients are asked to indicate their levels of belief frequency with a 5-level scale (0-4: 0 indicates not at all and 3 all the time) at 13 questions. A sum of all responses is calculated (52 being the maximum) for analysis. The higher the value the higher the levels of catastrophizing.
Kinesiophobia | 3 months
  Kinesiophobia will be assessed with the Tampa Scale for Kinesiophobia (TSK) where patients are asked to indicate their levels of agreement with a 4-level scale (1-4: 1 indicates not at all and 3 all the time) at 17 questions. A sum of all responses is calculated (68 being the maximum) for analysis. The higher the value the higher the levels of kinesiophobia.
Neuropathic Pain: Pain-DETECT questionnaire (PD-Q) | 3 months
  Neuropathic pain will be assessed with the Pain-DETECT questionnaire (PD-Q) where patients are firstly asked to describe the course of their pain by choosing one of 3 different pictures. A value has been allocated to each picture (-1, 0, +1 and +1). Secondly they are asked to indicate (yes or no) whether their pain radiates to a different part of their body. Yes is marked with +2 whereas No with 0. Thirdly, patients are asked to indicate their symptom intensity with a 6-level scale (0-5: 0 indicates never and 5 very strongly) at 7 questions. A sum of all responses is calculated and a final value is formed with the addition of the values from step one and two (38 being the maximum) for analysis. The higher the value the higher the levels of neuropathic pain.
Widespread Pain | 3 months
  Widespread pain will be assessed with the the use of a blank body manikin where patients are asked to draw the areas of pain on the manikin. Unbeknownst to patients, the manikin is divided into 46 body areas. A categorical variable is entered (1 for pain on the area, 0 for no pain) according to the pain distribution of the patients. No single value can be produced for analysis. Areas distant to the primary area of pain (Lower Back), like the chest or the forearm, will be used as independent variables in a multivariate regression model.
Fibromyalgia Severity | 3 months
  Fibromyalgia severity will be assessed with the Fibromyalgia Severity Scale (FMSS) where patients are firstly asked to tick a box on a body manikin if they feel pain on that area. Each tick is marked with 1 point. Then, patients are asked to indicate their symptom severity with a 4-level scale (0-3: 0 = no problem and 3 = severe) at 3 questions about tiredness, sleep and forgetfulness. A sum of all responses is calculated and is added to the total manikin value. Lastly, patients are asked to indicate whether they experienced headaches, depression and abdominal pain amongst 37 other symptoms. If they did, a point for each symptom is added on their overall mark (min: 0, max: 31). The higher the overall value the higher the severity of fibromyalgia.
Health care utilisation | 3 months
  Health care utilisation will be measured with the unvalidated Health Care Utilisation Questionnaire for Low Back Pain (HCUQ-LBP) where patients will be asked to indicate the type and amount of health care utilisation (visits to hospital, visits/calls to general practitioners (GPs) and practice nurses, use of social care, physiotherapists, chiropractors, psychologists, osteopaths and occupational therapists) in the last 3 months. Every health care use will be marked with a point and a total value will be produced for analysis (min: 0, max: any). The higher the value the higher the health care utilisation.
Medication type utilisation | 3 months
  Medication type utilisation will be determined when patients will be asked to record on a specially designed sheet the type of received medication in the last three months. Separate categories will be formed according to medication type (e.g. anti-inflammatory non-steroidal drugs, steroids, opioids, non-opioids) and a categorical variable will be stored (1 for yes, 0 for no) on these categories. No single value can be produced for analysis for this sub-questionnaire. Categories of medication types will be used as categorical independent variables in a multivariate regression model.

OTHER OUTCOMES:
Course of low back pain: Keele Stratification and Screening Tool for Low Back Pain (STarT-Back) | 3 months
  The prognosis of Low Back Pain will be determined with the Keele Stratification and Screening Tool for Low Back Pain (STarT-Back) where patients are asked to agree or disagree with 8 sentences (tick appropriately) and on a 9th question indicate how bothersome their back pain is on a 5-level scale (not at all to extremely). Every agreement is marked with 1 point as well as if patients rate their back pain as very much or extremely bothersome. A sum of all responses is calculated (9 being the maximum) for interpretation and analysis. The higher the value the higher the risk of unfavourable prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Walsh, Principal Investigator — The University of Nottingham
Locations (1):
- King's Mill Hospital, Sutton in Ashfield, Nittinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manusov EG. Evaluation and diagnosis of low back pain. Prim Care. 2012 Sep;39(3):471-9. doi: 10.1016/j.pop.2012.06.003. PMID 22958556
- [Background] Ramond A, Bouton C, Richard I, Roquelaure Y, Baufreton C, Legrand E, Huez JF. Psychosocial risk factors for chronic low back pain in primary care--a systematic review. Fam Pract. 2011 Feb;28(1):12-21. doi: 10.1093/fampra/cmq072. Epub 2010 Sep 10. PMID 20833704
- [Background] Bridges, S., Chronic Pain, in Health Survey for England 2011. 2012, Health and Social Care Information Centre: UK.
- [Background] May S. Self-management of chronic low back pain and osteoarthritis. Nat Rev Rheumatol. 2010 Apr;6(4):199-209. doi: 10.1038/nrrheum.2010.26. PMID 20357789
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] de Silva, D., Helping people help themselves: A review of the evidence considering whether it is worthwhile to support self-management. 2011: Health Foundation.
- [Background] Du S, Hu L, Dong J, Xu G, Chen X, Jin S, Zhang H, Yin H. Self-management program for chronic low back pain: A systematic review and meta-analysis. Patient Educ Couns. 2017 Jan;100(1):37-49. doi: 10.1016/j.pec.2016.07.029. Epub 2016 Jul 25. PMID 27554077
- [Background] O'Sullivan, P., et al., Multidimesional approach for the targeted management of low back pain, in Grieve's Modern Musculoskeletal Physiotherapy: Vertebral Column and Peripheral Joints, G. Jull, et al., Editors. 2015, Elsevier Health Sciences: UK. p. 465-470.
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Background] Smart KM, Blake C, Staines A, Doody C. Self-reported pain severity, quality of life, disability, anxiety and depression in patients classified with 'nociceptive', 'peripheral neuropathic' and 'central sensitisation' pain. The discriminant validity of mechanisms-based classifications of low back (+/-leg) pain. Man Ther. 2012 Apr;17(2):119-25. doi: 10.1016/j.math.2011.10.002. Epub 2011 Nov 9. PMID 22074733
- [Background] Panagioti M, Richardson G, Small N, Murray E, Rogers A, Kennedy A, Newman S, Bower P. Self-management support interventions to reduce health care utilisation without compromising outcomes: a systematic review and meta-analysis. BMC Health Serv Res. 2014 Aug 27;14:356. doi: 10.1186/1472-6963-14-356. PMID 25164529
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] Nijs J, Van Oosterwijck J, De Hertogh W. Rehabilitation of chronic whiplash: treatment of cervical dysfunctions or chronic pain syndrome? Clin Rheumatol. 2009 Mar;28(3):243-51. doi: 10.1007/s10067-008-1083-x. Epub 2009 Jan 22. PMID 19160000
- [Background] Jull G, Sterling M, Kenardy J, Beller E. Does the presence of sensory hypersensitivity influence outcomes of physical rehabilitation for chronic whiplash?--A preliminary RCT. Pain. 2007 May;129(1-2):28-34. doi: 10.1016/j.pain.2006.09.030. Epub 2007 Jan 10. PMID 17218057
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Murphy SL, Lyden AK, Phillips K, Clauw DJ, Williams DA. Subgroups of older adults with osteoarthritis based upon differing comorbid symptom presentations and potential underlying pain mechanisms. Arthritis Res Ther. 2011 Aug 24;13(4):R135. doi: 10.1186/ar3449. PMID 21864381
- [Background] Nijs, J., et al., The neurophysiology of pain and pain modulation: Modern pain neuroscience for musculoskeletal physiotherapists, in Grieve's Modern Musculoskeletal Physiotherapy: Vertebral Column and Peripheral Joints, G. Jull, et al., Editors. 2015, Elsevier Health Sciences: UK.
- [Background] Geber C, Klein T, Azad S, Birklein F, Gierthmuhlen J, Huge V, Lauchart M, Nitzsche D, Stengel M, Valet M, Baron R, Maier C, Tolle T, Treede RD. Test-retest and interobserver reliability of quantitative sensory testing according to the protocol of the German Research Network on Neuropathic Pain (DFNS): a multi-centre study. Pain. 2011 Mar;152(3):548-556. doi: 10.1016/j.pain.2010.11.013. Epub 2011 Jan 14. PMID 21237569
- [Background] Pfau DB, Krumova EK, Treede RD, Baron R, Toelle T, Birklein F, Eich W, Geber C, Gerhardt A, Weiss T, Magerl W, Maier C. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): reference data for the trunk and application in patients with chronic postherpetic neuralgia. Pain. 2014 May;155(5):1002-1015. doi: 10.1016/j.pain.2014.02.004. Epub 2014 Feb 10. PMID 24525274
- [Background] Sterling M, Jull G, Vicenzino B, Kenardy J, Darnell R. Physical and psychological factors predict outcome following whiplash injury. Pain. 2005 Mar;114(1-2):141-8. doi: 10.1016/j.pain.2004.12.005. Epub 2005 Jan 21. PMID 15733639
- [Background] Backonja MM, Attal N, Baron R, Bouhassira D, Drangholt M, Dyck PJ, Edwards RR, Freeman R, Gracely R, Haanpaa MH, Hansson P, Hatem SM, Krumova EK, Jensen TS, Maier C, Mick G, Rice AS, Rolke R, Treede RD, Serra J, Toelle T, Tugnoli V, Walk D, Walalce MS, Ware M, Yarnitsky D, Ziegler D. Value of quantitative sensory testing in neurological and pain disorders: NeuPSIG consensus. Pain. 2013 Sep;154(9):1807-1819. doi: 10.1016/j.pain.2013.05.047. Epub 2013 Jun 3. PMID 23742795
- [Background] Uddin Z, MacDermid JC, Galea V, Gross AR, Pierrynowski MR. The current perception threshold test differentiates categories of mechanical neck disorder. J Orthop Sports Phys Ther. 2014 Jul;44(7):532-40, C1. doi: 10.2519/jospt.2014.4691. PMID 24981222
- [Background] Cruccu G, Anand P, Attal N, Garcia-Larrea L, Haanpaa M, Jorum E, Serra J, Jensen TS. EFNS guidelines on neuropathic pain assessment. Eur J Neurol. 2004 Mar;11(3):153-62. doi: 10.1111/j.1468-1331.2004.00791.x. PMID 15009162
- [Background] Hill JC, Dunn KM, Lewis M, Mullis R, Main CJ, Foster NE, Hay EM. A primary care back pain screening tool: identifying patient subgroups for initial treatment. Arthritis Rheum. 2008 May 15;59(5):632-41. doi: 10.1002/art.23563. PMID 18438893
- [Background] Traeger A, McAuley JH. STarT Back Screening Tool. J Physiother. 2013 Jun;59(2):131. doi: 10.1016/S1836-9553(13)70170-X. No abstract available. PMID 23663803
- [Background] Hill JC, Whitehurst DG, Lewis M, Bryan S, Dunn KM, Foster NE, Konstantinou K, Main CJ, Mason E, Somerville S, Sowden G, Vohora K, Hay EM. Comparison of stratified primary care management for low back pain with current best practice (STarT Back): a randomised controlled trial. Lancet. 2011 Oct 29;378(9802):1560-71. doi: 10.1016/S0140-6736(11)60937-9. Epub 2011 Sep 28. PMID 21963002
- [Background] Knofczynski, G.T. and D. Mundfrom, Sample sizes when using multiple linear regression for prediction. Educational and Psychological Measurement, 2008. 68(3): p. 431-442.